CLINICAL TRIAL: NCT06331949
Title: The Effect of Video-Assisted Training Given to Pregnant Women on Non-Stress Test Application on Pregnancy Stress and Prenatal Attachment
Brief Title: Video Supported Training on Non-Stress Test Application to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Özbek (Other)
Responsible Party: Sponsor-Investigator, Hilal Özbek, Assist. Prof. Dr., Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TR TOKAT02
Record Dates: First submitted 2024-03-16; First posted 2024-03-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: First Pregnancy
Keywords: NST; prenatal attachment; video; education; State-Trait Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to midwifery care, training content, training videos and brochure-supported training on NST will be provided. The NST device will be inserted and, to be standard, 5 minutes after the procedure begins, the volume of the fetal heart sound coming from the device will be increased during the NST recording and the fetal heart sound will be ensured to continue. The pregnant woman who will be transferred will rest for about 2 minutes.
  Interventions: Other: video assisted training
- Control Group (No Intervention): No additional applications will be made

INTERVENTIONS:
Other: video assisted training — Ebelik bakımının yanı sıra NST konusunda eğitim içerikleri, eğitim videoları ve broşür destekli eğitimler verilecek. NST cihazı takılacak ve standart olarak işlem başladıktan 5 dakika sonra NST kaydı sırasında cihazdan gelen fetal kalp sesinin şiddeti artırılarak fetal kalp sesinin devam etmesi sağlanacaktır. Transfer edilecek hamile kadın yaklaşık 2 dakika kadar dinlenecektir.
  Arms: Experimental Group

SUMMARY:
Women go through many practices during their pregnancy. These practices, along with ignorance, create stress in the mother. However, performing the procedures for the first time may increase the mother's stress level. Stress during pregnancy also affects prenatal attachment. Non-Stress Test (NST) Application is a test applied to pregnant women starting from the 28th week of pregnancy and provides information about the baby's well-being and uterine contractions. There is a gap in the literature regarding education for pregnant women undergoing NST regarding stress levels and prenatal attachment. With this study, stress levels and prenatal attachment levels in pregnant women will be determined during NST, which is frequently applied during pregnancy. Additionally, the effects of midwifery care in this process will be realized. In this way, solutions will be produced for problems that may arise. A better quality of midwifery care will be provided

DETAILED DESCRIPTION:
Background: NST may negatively affect the stress level and prenatal attachment level in primiparous pregnant women.

Purpose: This study will be carried out to determine the effect of video-educated midwifery care given to primiparous pregnant women before NST application on pregnancy stress and prenatal attachment levels.

Method: The data of the research will be collected at Tokat State Hospital after permission. During data collection, pregnant women who apply to the NST room of the relevant hospital and meet the inclusion criteria for the study will be informed about the researchers and the study. Written consent will be obtained from pregnant women who volunteer to participate in the study by filling out the "Informed Volunteer Consent Form". The training will be held in a suitable room (a quiet room where individuals can sit comfortably and see each other) in the area where the NST room is located in the hospital. Pregnant women will be informed about the purpose of the study, the confidentiality of the answers, where and how the data will be stored, and their questions on the subject will be answered. Data collection forms will be given to the participant by the researcher and they will be asked to fill them out. The data collection forms will be checked by the researcher to see if they have been filled out completely. This process is planned to take approximately 10-15 minutes.

Experimental Group: In addition to midwifery care, training content, training videos and brochure-supported training on NST will be provided. The NST device will be inserted and, to be standard, 5 minutes after the procedure begins, the volume of the fetal heart sound coming from the device will be increased during the NST recording and the fetal heart sound will be ensured to continue. The pregnant woman who will be transferred will rest for about 2 minutes.

Control Group: No additional applications will be made

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant woman
* Able to read and write
* Pregnant women who are 32 weeks or more pregnant
* No detection problems
* The baby has no health problems
* Having no psychological or physiological health problems
* Pregnant women who accept the research

Exclusion Criteria:

* Under 32 weeks
* Those who did not accept the research
* If the pregnant woman feels uncomfortable during the research,
* Pregnant women who want to leave any part of the research

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | Baseline]
  It requires the person to mark one of four options, such as 1 (Not at all), 2 (Somewhat), 3 (A lot), 4 (Completely), depending on the intensity of his/her feelings about himself/herself at a certain time and under certain conditions.
Prenatal Attachment Inventory (PAI) | Baseline]
  PAI is used to explain the thoughts, feelings, and situations experienced by the woman during pregnancy and to determine the level of attachment to the baby in the prenatal period. The increase in the score received by the pregnant woman indicates that her attachment level also increases.

SECONDARY OUTCOMES:
State-Trait Anxiety Scale | after training is completed
  It requires the person to mark one of four options, such as 1 (Not at all), 2 (Somewhat), 3 (A lot), 4 (Completely), depending on the intensity of his/her feelings about himself/herself at a certain time and under certain conditions.
Prenatal Attachment Inventory (PAI) | after training is completed
  PAI is used to explain the thoughts, feelings, and situations experienced by the woman during pregnancy and to determine the level of attachment to the baby in the prenatal period. The increase in the score received by the pregnant woman indicates that her attachment level also increases.

OTHER OUTCOMES:
State-Trait Anxiety Scale | two weeks after training is completed
  It requires the person to mark one of four options, such as 1 (Not at all), 2 (Somewhat), 3 (A lot), 4 (Completely), depending on the intensity of his/her feelings about himself/herself at a certain time and under certain conditions.
Prenatal Attachment Inventory (PAI) | two weeks after training is completed
  PAI is used to explain the thoughts, feelings, and situations experienced by the woman during pregnancy and to determine the level of attachment to the baby in the prenatal period. The increase in the score received by the pregnant woman indicates that her attachment level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Özbek, Principal Investigator — Tokat Gaziosmanpasa Universty; Nil Şevval Demir, Student, Principal Investigator — Tokat Gaziosmanpasa Universty
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya, D. (2021). Gebeliğin Oluşumu ve Fizyolojisi. Içinde Ö. Doğan Yüksekol, F. Evcili, & G. Doğaner (Ed.), Normal gebelik ve bakım (1. bs, ss. 64-86). Ankara Nobel Tıp Kitapevleri.
- [Background] Aksay, Y., Gülhan, Y. B., Saygın, N., & Körükçü, Ö. (2017). Gebelerin Psikososyal Sağlıkları Doğum Tercihini Etkiler Mi? Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi, 6(4), 138-145
- [Background] Kaloğlu Bi̇ni̇ci̇, D., & Köse Tuncer, S. (2020). Primipar ve Multipar Gebelerde Algılanan Stres ve Etkileyen Faktörlerin İncelenmesi. Ebelik ve Sağlık Bilimleri Dergisi, 3(3), 189-202.
- [Background] Özkan, H., & Mucuk, Ö. (2021). Gebelikte Ruh Sağlığında Meydana Gelen Değişimler ve Bakım. Içinde Ö. Doğan Yüksekol, F. Evcili, & G. Doğaner (Ed.), Normal gebelik ve bakım (1. bs, ss. 175-184). Ankara Nobel Tıp Kitapevleri.
- [Background] Genç Koyucu, R., Ülkar, D., & Erdem, B. (2020). Primipar ve Multipar Gebelerin Gebelik Streslerinin Karşılaştırılması. İnönü Üniversitesi Sağlık Hizmetleri Meslek Yüksekokulu Dergisi, 8(3), 652-663. https://doi.org/10.33715/inonusaglik.745511
- [Background] Nakamura Y, Okada T, Morikawa M, Yamauchi A, Sato M, Ando M, Ozaki N. Perinatal depression and anxiety of primipara is higher than that of multipara in Japanese women. Sci Rep. 2020 Oct 13;10(1):17060. doi: 10.1038/s41598-020-74088-8. PMID 33051530
- [Background] Üst, Z. D., & Pasinlioğlu, T. (2015). Primipar ve Multipar Gebelerde Doğum ve Postpartum Döneme İlişkin Endişelerin Belirlenmesi. Journal of Health Science and Profession, 2(3), 306-317. https://doi.org/10.17681/HSP.96963
- [Background] Bakır, N., & Sarızayim, Ş. (2020). The relationship between psychosocial health and prenatal attachment in pregnant women. Perinatal Journal , 28(2), 73-81. https://doi.org/10.2399/prn.20.0282006
- [Background] Karakas NM, Dagli FS. The importance of attachment in infant and influencing factors. Turk Pediatri Ars. 2019 Jul 11;54(2):76-81. doi: 10.14744/TurkPediatriArs.2018.80269. eCollection 2019. PMID 31384141
- [Background] McNamara J, Townsend ML, Herbert JS. A systemic review of maternal wellbeing and its relationship with maternal fetal attachment and early postpartum bonding. PLoS One. 2019 Jul 25;14(7):e0220032. doi: 10.1371/journal.pone.0220032. eCollection 2019. PMID 31344070
- [Background] Alan Dikmen, H., & Çankaya, S. (2018). Maternal Obezitenin Prenatal Bağlanma Üzerine Etkisi. Acibadem Universitesi Saglik Bilimleri Dergisi, 9(2), 118-123. https://doi.org/10.31067/0.2018.1
- [Background] Alkaş, Ü., & Varışoğlu, Y. (2023). Primipar Gebelerde Anksiyete ve Prenatal Bağlanma: Pandemi Sürecinin Etkileri. Journal of Women's Health Nursing Jowhen , 9(1), 1-11. https://dergipark.org.tr/en/pub/kashed/issue/76497/1203330
- [Background] Bilgin, Z., & Ecevit Alpar, Ş. (2018). Kadınların Maternal Bağlanma Algısı ve Anneliğe İlişkin Görüşleri . Journal of Health Science and Profession, 5(1), 6-15. https://doi.org/10.17681/HSP.296664
- [Background] Şimşek, H. N., & Bolsoy, N. (2018). Düzce Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi " Gönderim " Sosyal Destek Sistemleri ve Ebelik. Düzce Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi, 8(2), 97-103. https://dergipark.org.tr/en/pub/duzcesbed/issue/37762/338959?publisher=duzce
- [Background] Kınık, E., & Özcan, H. (2020). Maternal Bağlanmayı Etkileyen Faktörler ve Primiparlarda Maternal Bağlanma Durumu. Journal of Health Profession Research, 2(1), 47-53. https://dergipark.org.tr/en/pub/jhpr/issue/52597/596869
- [Background] Aktulay, A., Üstün, Y. E., Eyi, E. G. Y., Yörük, Ö., Hançerlioğulları, N., & Mollamahmutoğlu, L. (2013). Nonreaktif Nst Ön Tanısının Düşük Riskli Gebeliklerde Değerlendirilmesi. Jinekoloji-Obstetrik ve Neonatoloji Tıp Dergisi, 10(37), 1542-1545. https://dergipark.org.tr/en/pub/jgon/issue/51917/676229
- [Background] Kuru İyidir, Z. (2021). Non-Stress Teste Yönelik Verilen Eğitimin Gebelerin Kaygı Düzeyine Etkisi [Yüksek Lisans Tezi]. Aydın Adnan Menderes Üniversitesi Sağlık Bilimleri Enstitüsü.
- [Background] Çoban, M. (2022). Non Stres Test Esnasında Sanal Gözlük Kullanımının Kaygı, Stres Ve Fetal İyilik Üzerine Etkisi. [Yüksek Lisans Tezi]. İnönü Üniversitesi Sağlık Bilimleri Fakültesi.
- [Background] Hoca Nacar, E., & Gökkaya, F. (2019). Bağlanma ve Maternal Bağlanma Konusunda Bir Derleme. Cyprus Turkish Journal of Psychiatry and Psychology, 1(1), 49-55. https://doi.org/10.35365/ctjpp.19.1.06
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Cohen, J. (1988). The t test for means. Statistical Power Analysis For the Behavioural Sciences . (N. Hillsdale, Ed.; 2. bs).
- [Background] Polit, D., & Beck, C. (2017). Nursing research: Generating and assessing evidence for nursing practice (10th ed.). PA: Lippincott Williams & Wilkins.